CLINICAL TRIAL: NCT03606564
Title: Parent's Perception and Compliance With Pre-operative Fasting Instructions in Paediatric Patients Undergoing Day Care Surgery
Brief Title: Parents Perception and Compliance With Pre Operative Fasting Instructions in Paediatric Patients
Status: Completed | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, KARAN SINGLA, Principal Investigator, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: 9605/PG-2Trg/2013/13402
Record Dates: First submitted 2018-05-31; First posted 2018-07-31 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Fasting
Keywords: compliance; fasting guidelines
MeSH Terms: conditions — Fasting; Patient Compliance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- paediatric patients undergoing day care surgery
  Interventions: Other: study of fasting time among pediatric patients undergoing day care surgery

INTERVENTIONS:
Other: study of fasting time among pediatric patients undergoing day care surgery — parents of children undergoing day care surgery were given a questionnaire to be filled containing questions regarding time of fasting that was instructed and

SUMMARY:
This study evaluates the perception and compliance with the fasting instructions given to parents of children undergoing surgery. A questionnaire was provided to the parents indicating fasting time requested and actual time of fasting.

DETAILED DESCRIPTION:
American Society of Anesthesiologists (ASA) have recommended fasting guidelines of 8 hours of solids, 6 hours for formula milk, 4 hours for breast milk and 2 hours of clear liquids, for preoperative patients undergoing elective surgery. Parents of Children undergoing surgery are instructed to adhere to these guidelines. Parents might not be compliant with these instructions. They may fast their children less than or more than the recommended time.

Main aim of this study is to find out the incidence of non compliance with the fasting instructions and try to find the reasons for such non compliance.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 to 12 years
* ASA I and II category
* Elective day care surgery
* General anaesthesia planned

Exclusion Criteria

* Parent's refusal to participate.
* Children with complex nutritional requirements eg. feeding via gastrostomy tube
* Parents who cannot read or understand English, Hindi or Punjabi

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Consecutive children aged 1 to 12 years of ASA I and II category, scheduled to undergo elective day care surgery under general anaesthesia, were included in this prospective study
Sampling Method: Probability Sample
Enrollment: 1050 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Median duration of fasting | 1.5 years
  Median time of pre operative fasting as advised by anaesthesiologist/surgeon/nurse in the Pre Anaesthesia Clinic was compared with the Median duration of fasting of the patient just before surgery.
Percentage of parents who followed the preoperative fasting instructions | 1.5 years
  Percentage of parents who adhered to advised fasting time was compared with percentage of parents who fasted their children more than or less than what was advised.

SECONDARY OUTCOMES:
Percentage of parents who attended Pre Anaesthesia Clinic | 1.5 years
Percentage of parents who could recall fasting instructions that were provided in Pre Anaesthesia Clinic | 1.5 years
Percentage of parents who could tell if they were provided separate fasting instructions for solids and liquid foods | 1.5 years
Percentage of parents who could recall if fasting instructions were verbal or written orders | 1.5 years
Percentage of parents who received fasting instructions from anyone other than the anaesthetist | 1.5 years
Percentage of parents who understood the actual reason to fast before surgery | 1.5 years
Percentage of patients who were not adequately fasted. | 1.5 years
Percentage of parents who complained about fasting time being too long for their children | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: indu bala, MD, Principal Investigator — PGIMER, chandigarh, india
Locations (1):
- Post Graduate Institute of Medical Education and Research,, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No